CLINICAL TRIAL: NCT05007184
Title: Evaluating Food Policy Interventions Using NUSMart
Brief Title: Understanding Food Choices in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: World Bank (Other); Public Health Authority of Saudi Arabia (Unknown)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 7197919
Record Dates: First submitted 2021-08-03; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Diet Quality
Keywords: front-of-pack labels; online grocery shopping; Kingdom of Saudi Arabia; Chilean warning labels; Nutri-Score labels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Arm 1) (No Intervention): Participants will experience an unmodified version of NUSMart, which replicates the traditional shopping experience of online grocery stores.
- Warning Label Arm (Arm 2) (Experimental): Similar to Arm 1 except that products are labeled with Chilean warning FOP labels.
  Interventions: Behavioral: Chilean Warning Labels
- Nutri-Score Arm (Arm 3) (Experimental): Similar to Arm 1 except that products are labeled with NutriScore FOP labels.
  Interventions: Behavioral: Nutri-Score Labels

INTERVENTIONS:
Behavioral: Chilean Warning Labels — These labels were implemented in Chile in 2016. They are shown on those less-healthy food and beverage products that do not fall within thresholds that are defined for the following nutrients: sugar, sodium, calories and saturated fats. The original labels are in Spanish but the ones that we displayed were in Arabic.
  Arms: Warning Label Arm (Arm 2)
Behavioral: Nutri-Score Labels — These labels were implemented by the French government in 2017. They are shown on all food and beverage products and range from A to E with the corresponding colours moving from Green to Red (symbolizing best to worst). The scores and grades are calculated based on 7 different nutrients grouped into 2 categories i.e. nutrients to consume (such as fibre) and nutrients to avoid (such as sugar). We modified the labels by adding % sugar per serving on the right side of the labels.
  Arms: Nutri-Score Arm (Arm 3)

SUMMARY:
Using a 3-arm randomized controlled trial, the investigators aim to rigorously evaluate the effects of two front-of-pack (FOP) food labels on diet quality. The first food label is a modified version of Chilean warning FOP label and the second food label is a modified version of French FOP label, Nutri-Score. The investigators used an experimental online grocery store, called NUSMart, which is similar in design to commercial web-based grocery stores to test these two FOP labels. Participants were randomly assigned to one of the following arms and asked to complete a one-time hypothetical shop.

Arm 1: Participants experienced a default version of NUSMart which replicated the traditional shopping experience of online grocery stores with no FOP labels (Control).

Arm 2: Same as Arm 1 NUSMart except that Chilean warning FOP labels were displayed on less healthy food and beverages. Products with specific nutrients (i.e. sugar, sodium, saturated fat, energy) falling outside the bounds of the thresholds defined by the Chilean warning labels were depicted with the warning labels on them.

Arm 3: Same as Arm 1 NUSMart except that Nutri-Score FOP labels along with % sugar per serving were displayed on all food and beverages. These labels score products on the basis of 7 nutrients (calories, saturated fats, sugar, salt, fibre, protein and percentage of fruits, vegetables and nuts) from A to E (best to worst). To ensure that participants understood what Nutri-Score labels mean and how they work, an introductory video was shown before shopping.

The investigators hypothesize the following:

Hypothesis 1: Diet quality, as measured by weighted average Nutri-Score point of shoppers' final baskets, will be greatest in Arm 3, followed by Arm 2, followed by Control.

Hypothesis 2: Grams of sugar per serving/ milligrams of sodium per serving/ grams of saturated fat per serving/ calories per serving will be least in Arm 2, followed by Arm 3, followed by Control.

DETAILED DESCRIPTION:
Experimental design & procedures

The aim of this study is to use a 3-arm randomized controlled trial with an online grocery store (NUSMart), to rigorously evaluate the effect of the two FOP labels, Chilean warning labels and Nutri-Score, on diet quality.

1. Food labels

   The investigators tested 2 different types of food labels in this study. They are as follows:
   1. Chilean Warning Labels: These labels were implemented in Chile in 2016. They are shown on those less-healthy food and beverage products that don't fall within thresholds that are defined for the following nutrients: sugar, sodium, calories and saturated fats. The original labels are in Spanish but the ones that the investigators displayed were in Arabic.
   2. Nutri-Score Labels: These labels were implemented by the French government in 2017. They are shown on all food and beverage products and range from A to E with the corresponding colours moving from Green to Red (symbolizing best to worst). The scores and grades are calculated based on 7 different nutrients grouped into 2 categories i.e. nutrients to consume (such as fibre) and nutrients to avoid (such as sugar). The investigators modified the labels by adding % sugar per serving on the right side of the labels.
2. Overview of RCT Design

   To test these labels, the investigators used three different versions of NUSMart. Each participant was randomly assigned to one of the following arms and asked to complete a one-time hypothetical shop.

   Arm 1: Control arm. Participants experienced an unmodified version of NUSMart, which replicates the traditional shopping experience of online grocery stores.

   Arm 2: Similar to Arm 1 except that products were labeled with Chilean warning FOP labels.

   Arm 3: Similar to Arm 1 except that products were labeled with NutriScore FOP labels.

   To minimize hypothetical shopping biases, the investigators set a minimum spending value per person per week and adjusted the total minimum spending value depending on household size.
3. Subject related procedures

As the investigators have done in prior studies, participants were recruited if they were KSA residents aged 18 years or older, could speak Arabic and were primary weekly shoppers for their households. Recruitment was done using a Saudi Arabia based web panelist.

On recruitment, they were asked to fill in a baseline questionnaire to collect demographic and health characteristics, which took approximately 10-15 minutes to complete.

The baseline questionnaire includes a question as to whether any household members have a medical condition, such as diabetes or hypertension, which requires limiting the types of foods they eat. The investigators asked this question to allow for testing whether the interventions differentially influence these households, with the expectation that households with less healthy patients may obtain greater benefits from purchasing baskets with higher mean Nutri-Scores. Since the objective of this RCT is to quantify the effectiveness of the interventions on diet quality, a precursor to NCDs, the collection of household health indicators is reasonable.

Upon completion of the baseline survey, participants were randomly assigned to one of the 3 shopping conditions (Arm 1 [Control], Arm 2, or Arm 3). They logged into the NUSMart website and were asked to purchase their weekly groceries with a minimum spend per person per week (the total minimum spending value depends on the household size). Each participant therefore shopped only once during the study in one of the arms (1,2 or 3) which was randomly assigned to them.

Participants were given explicit instructions to purchase groceries for the purposes of breakfast, lunch, dinner, snacks and beverage consumption for one week keeping in mind that they would not be consuming any meals outside. The stores were set up such that participants were not allowed to check out with their cart unless they selected items from at least 4 different NUSMart categories. This ensures that participants shop as though they are shopping for their own consumption i.e. to minimize hypothetical biases.

A post-study survey was conducted after the last shop to collect participant opinions on the labels and understand their impact better.

ELIGIBILITY:
Inclusion Criteria:

* People who are KSA (Kingdom of Saudi Arabia) citizens
* Age of 18 and above,
* Arabic speakers, and
* A weekly primary grocery shopper for their households can participate in this study.

Exclusion Criteria:

* People who are not KSA citizens,
* Under 18 years of age,
* Cannot speak Arabic, or
* Are not weekly primary grocery shoppers for their households cannot participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Value of Nutri-Score | After completion of data collection, an average of about 1 month
  Diet quality measured by the weighted average of all purchased products' Nutri-Score for the shopping trip. Nutri-Score is an individual dietary index based on the British Food Standard Agency Nutrient Profiling System.

SECONDARY OUTCOMES:
Quantity of other Nutrients | After completion of data collection, an average of about 1 month
  grams of sugars per serving/ milligrams of sodium per serving/ grams of saturated fat per serving/ calories per serving.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No